CLINICAL TRIAL: NCT05309161
Title: Efficacy Testing of Crassocephalum Rabens Extract Capsules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Greenyn Biotechnology Co., Ltd. (Industry)
Collaborators: Chia Nan University of Pharmacy ＆ Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-129-A
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-03

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (placebo) (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Crassocephalum rabens extract
- B group (experimental) (Active Comparator): Crassocephalum rabens extract
  Interventions: Dietary Supplement: Crassocephalum rabens extract

INTERVENTIONS:
Dietary Supplement: Crassocephalum rabens extract — dosage: a capsule (180 mg)/day; duration: 1 month

SUMMARY:
This study is to investigate the improveing effects of the Crassocephalum rebens extract on skin conditions in normal people.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 20 years
2. Healthy people

Exclusion Criteria:

1. Non-volunteer
2. Pregnant and lactating women
3. Hypersensitivity to the assigned product
4. Diagnosed with skin diseases, liver diseases, kinedy disease, and other severe diseases
5. Cosmetic, drug, or food allergies
6. Concurrent aesthetic treatments (e.g., intense pulse light, medical peelings, or laser therapy)
7. Aceepted aesthetic treatments one month ago before the study
8. Chronic sun exposure (over 3 hours/day)
9. The members of the research team

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Measurement of skin hydration | Week 0
  Corneometer CM825 is used to measure the moisture of upper cheek (unit: Corneometer® unit)
Measurement of skin hydration | Week 4
  Corneometer CM825 is used to measure the moisture of upper cheek (unit: Corneometer® unit)
Measurement of skin brightness | Week 0
  Chroma Meter MM500 is employed to measure the brightness of upper cheek (unit: L* value (L* range: 0-100)).
Measurement of skin brightness | Week 4
  Chroma Meter MM500 is employed to measure the brightness of upper cheek (unit: L* value (L* range: 0-100)).
Measurement of skin texture | Week 0
  Visia® skin analysis system is used to measure the skin texture of full face (unit: number of fine lines)
Measurement of skin texture | Week 4
  Visia® skin analysis system is used to measure the skin texture of full face (unit: number of fine lines)
Measurement of skin spots | Week 0
  Visia® skin analysis system is used to measure the skin spots of full face (unit: number of spots)
Measurement of skin spots | Week 4
  Visia® skin analysis system is used to measure the skin spots of full face (unit: number of spots)
Measurement of collagen content | Week 0
  DermaLab® Series SkinLab Combo (Cortex) is employed to measure skin collagen content of upper cheek (unit: collagen density)
Measurement of collagen content | Week 4
  DermaLab® Series SkinLab Combo (Cortex) is employed to measure skin collagen content of upper cheek (unit: collagen density)
Measurement of Crow's feet | Week 0
  Visia® skin analysis system is used to measure the skin spots of full face (unit: number of Visia® skin analysis system is used to measure the skin spots of full face (unit: number of fine lines around eyes)
Measurement of Crow's feet | Week 4
  Visia® skin analysis system is used to measure the skin spots of full face (unit: number of Visia® skin analysis system is used to measure the skin spots of full face (unit: number of fine lines around eyes)
Measurement of skin elasticity | Week 0
  Cutometer® is used to measure the skin elasticity of upper cheek (unit: mm)
Measurement of skin elasticity | Week 4
  Cutometer® is used to measure the skin elasticity of upper cheek (unit: mm)
Measurement of skin wrinkles | Week 0
  Visia® skin analysis system is used to measure the skin wrinkles of full face (unit: number of wrinkles)
Measurement of skin wrinkles | Weeks 4
  Visia® skin analysis system is used to measure the skin wrinkles of full face (unit: number of wrinkles)
Measurement of skin pores | Week 0
  Visia® skin analysis system is used to measure the skin spots of full face (unit: number of pores)
Measurement of skin pores | Week 4
  Visia® skin analysis system is used to measure the skin spots of full face (unit: number of pores)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Principal Investigator — Department of Cosmetic Science, Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No